CLINICAL TRIAL: NCT03187873
Title: Chamas for Change: Validating an Integrated Community-based Strategy of Peer Support in Pregnancy and Infancy in Kenya
Brief Title: Chamas for Change Validation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Moi University (Other)
Collaborators: University of Toronto (Other); Indiana University (Other); AbbVie (Industry); Grand Challenges Canada (Other)
Responsible Party: Principal Investigator, Astrid Christoffersen-Deb, Visiting Lecturer, Moi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MoiU1
Record Dates: First submitted 2017-05-31; First posted 2017-06-15 (Actual); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Pregnancy Related
Keywords: community participation; Maternal and child health; Kenya

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chama cha MamaToto (Experimental): Women attending chamas will meet twice per month, receive social and health education from CHVs and participate in a savings/loans program.
  Interventions: Behavioral: Chama cha MamaToto
- Control (No Intervention): The CHVs in the control group will be given refresher training on health roles they are supposed to play according to the standard MOH activities

INTERVENTIONS:
Behavioral: Chama cha MamaToto — Chamas are a community-led model of peer support for women in pregnancy and infancy. Chamas are highly gendered institutions that women have relied on for survival to pool resources. Using this existing cultural script, chamas have been tailored to the needs of pregnant women. Central to the approach is the integration of health, social and financial literacy education with a savings/loans program. Chamas are designed to improve MNCH by generating positive peer support for women to advocate for themselves and account for the care they receive.
  Arms: Chama cha MamaToto

SUMMARY:
This team has shown that chamas can be tailored to increase the uptake of health services in pregnancy and infancy, sustain themselves beyond the period of funding and become integrated within a county's health strategy. However, further investment is warranted to validate this intervention in a new region to ensure the positive effects on MNCH are a result of chamas and can be replicated. The purpose of this study is to demonstrate that chamas are an effective service-delivery platform for improving women's and children's health and well-being in western Kenya.

DETAILED DESCRIPTION:
The objectives are:

To test the effectiveness of chamas as an intervention on improving:

* Health services uptake (Facility delivery, attendance of 4 or more ANC visits, Visit by a CHV within 48 hours of birth, immunization uptake at 6 months-of-age, long-term FP uptake)
* Health behaviors and care practices (exclusive breastfeeding to 6 months)
* Women's Empowerment, peer support, parental stress, and harsh punishmennt within the home
* Maternal and infant morbidity (low birth weight, diarrhea in the last month, preterm deliveries)
* Maternal, perinatal, neonatal and infant mortality

To perform a qualitative evaluation to better understand women's and CHV's experience with chamas and understand how chamas affect peer support

To perform a process evaluation

To perform a cost effectiveness analysis on chamas.

The investigators plan to use a cluster randomized controlled design because the intervention is delivered in groups that are based within Community Units (CUs). We know that some of the positive effects of chamas expand to the community surrounding the chama. By randomizing clusters, we will hope to isolate these communities in order to understand the individual effects of chamas. The unit of randomization and implementation will be Community Units (CU). Because there are only 77 of the 163 CUs with active Community Health Workers trained by AMPATH, we will draw our intervention and control groups from these active units. By doing this, the control group is receiving the standard of care per the MOH and AMPATH community strategy. We will randomly assign each of the 77 active CUs in the four sub-counties to the chama intervention (arm 1) or to act as a control region (arm 2). We will evaluate individual outcomes on women enrolled in the study. The CUs that do not participate in the study will serve as buffer areas.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women < 28 weeks, and their newborn infants following birth

Exclusion Criteria:

-

Max Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3040 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Skilled Delivery | 1 year
  Proportion of women delivering in a health facility based on questionnaire

SECONDARY OUTCOMES:
Antenatal Care | 1 year
  Proportion of women attending 4 or more ANC visits based on questionnaire
Exclusive Breastfeeding | 17 months
  Proportion of women introducing solid foods after 6 months of age based on questionnaire
Contraception | 17 months
  Proportion of women initiating Long-Acting Reversible Contraception based on questionnaire
Health Insurance | 1 year
  Proportion of women with Health Insurance based on questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Christoffersen-deb, MDCM, Principal Investigator — Moi University; Julia Songok, MBChB, MMed, Principal Investigator — Moi University
Locations (1):
- Trans-Nzoia MOH Health Centers, Kitale, Trans Nzoia, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McHenry MS, Maldonado LY, Yang Z, Anusu G, Kaluhi E, Christoffersen-Deb A, Songok JJ, Ruhl LJ. Participation in a Community-Based Women's Health Education Program and At-Risk Child Development in Rural Kenya: Developmental Screening Questionnaire Results Analysis. Glob Health Sci Pract. 2021 Dec 21;9(4):818-831. doi: 10.9745/GHSP-D-20-00349. Print 2021 Dec 31. PMID 34933978
- [Derived] Maldonado LY, Bone J, Scanlon ML, Anusu G, Chelagat S, Jumah A, Ikemeri JE, Songok JJ, Christoffersen-Deb A, Ruhl LJ. Improving maternal, newborn and child health outcomes through a community-based women's health education program: a cluster randomised controlled trial in western Kenya. BMJ Glob Health. 2020 Dec;5(12):e003370. doi: 10.1136/bmjgh-2020-003370. PMID 33293295